CLINICAL TRIAL: NCT04570267
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Pharmacokinetics and Safety of Subcutaneous CSL324 in Healthy Japanese and White Subjects
Brief Title: Pharmacokinetics and Safety of Subcutaneous CSL324 in Healthy Japanese and White Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CSL324_1003
Record Dates: First submitted 2020-09-25; First posted 2020-09-30 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CSL324 (Low dose) (Experimental): One low dose of CSL324 administered subcutaneously on Day 1
  Interventions: Biological: CSL324
- CSL324 (High dose) (Experimental): One high dose of CSL324 administered subcutaneously on Day 1
  Interventions: Biological: CSL324
- Placebo (Placebo Comparator): One dose of placebo administered subcutaneously on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CSL324 — Sterile solution of recombinant anti G-CSF receptor monoclonal antibody for injection
  Other Names: Recombinant Anti G-CSF Receptor Monoclonal Antibody
  Arms: CSL324 (High dose); CSL324 (Low dose)
Drug: Placebo — Sterile solution of CSL324 formulation buffer for injection
  Arms: Placebo

SUMMARY:
Study CSL324_1003 is a single center, randomized, double-blind, placebo-controlled study designed to characterize and compare the PK properties and safety of a single subcutaneous dose of CSL324 in healthy Japanese and White subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female Japanese or White subjects aged 20 and 55 years, inclusive
* Body weight of at least 45 kg to 100 kg, inclusive
* Body mass index of 18.0 to 32.0 kg/m2, inclusive

Exclusion Criteria:

* A clinically significant medical condition, disorder, or disease of any organ system.
* Concurrent diagnosis of malignancy or history of malignancy (except for nonmelanoma skin cancer or cervical carcinoma in situ that has been adequately treated with no evidence of recurrence for at least 3 months before Screening).
* Immunosuppressive conditions and / or currently taking immunosuppressive or immunomodulative therapy.
* Clinically significant abnormalities on physical examination, vital signs, or laboratory assessments, or neutropenia (defined as absolute neutrophil count < 2.0 × 109/L).
* History of chronic or recurrent infections, clinical signs of active infection and / or fever, current / history of serious infection or hospitalized or received IV antibiotics for an infection in previous 2 months.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-12-09 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of CSL324 in serum | From Day 1 to Day 56
Area under the concentration-time curve from time 0 extrapolated to time infinity (AUC0-inf) of CSL324 in serum | From Day 1 to Day 56
Area under the concentration-time curve from time 0 to the last measurable concentration (AUC0-last) of CSL324 in serum | From Day 1 to Day 56

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events (TEAEs) by incidence, by severity, and by causality | Up to Day 56
Percentage of subjects with TEAEs by incidence, by severity, and by causality | Up to Day 56
Number of subjects with adverse events localized to the administration site by incidence, by severity, and by causality | Up to Day 7
Percentage of subjects with adverse events localized to the administration site by incidence, by severity, and by causality | Up to Day 7
Time to reach Cmax (Tmax) for CSL324 in serum | From Day 1 to Day 56
Terminal half-life (t1/2) for CSL324 in serum | From Day 1 to Day 56
Apparent clearance (CL/F) for CSL324 in serum | From Day 1 to Day 56
Apparent volume of distribution (Vz/F) for CSL324 in serum | From Day 1 to Day 56
Number of subjects with or without anti-CSL324 antibodies | Up to Day 56
Percentage of subjects with or without anti-CSL324 antibodies | Up to Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Scientia Clinical Research Ltd, Randwick, Australia

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider requests to share Individual Patient Data (IPD) from systematic review groups or bona-fide researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.
Supporting Information: Study Protocol, SAP
Time Frame: IPD requests may be submitted to CSL no earlier than 12 months after publication of the results of this study via an article made available on a public website.
Access Criteria: Requests may only be made by systematic review groups or bona-fide researchers whose proposed use of the IPD is non-commercial in nature and has been approved by an internal review committee.
  An IPD request will not be considered by CSL unless the proposed research question seeks to answer a significant and unknown medical science or patient care question as determined by CSL's internal review committee.
  The requesting party must execute an appropriate data sharing agreement before IPD will be made available.